CLINICAL TRIAL: NCT04860102
Title: Hands on vs Hands Off for Perineal Laceration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13/21
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Perineal Tear
MeSH Terms: interventions — Therapeutic Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hands on (Experimental): Hands-on was defined as involving one hand on the fetal head, applying pressure to control expulsion, with the other hand applying pressure on the maternal perineum
  Interventions: Procedure: hands on
- hands off (No Intervention): standard of care

INTERVENTIONS:
Procedure: hands on — Hands-on was defined as involving one hand on the fetal head, applying pressure to control expulsion, with the other hand applying pressure on the maternal perineum
  Arms: hands on

SUMMARY:
Perineal trauma at the time of vaginal delivery is common, and when the anal sphincter is included, these injuries can be associated with additional morbidity including incontinence, pelvic pain and sexual dysfunction. Techniques studied include hands-on vs hands-off, perineal massage, warm compresses, Ritgen maneuver, and others. It is unclear if a hands-on technique decreases the incidence of perineal trauma compared to a hands-off technique

DETAILED DESCRIPTION:
Different strategies have been adopted in the late first and/or second stage of labor to decrease the incidence of perineal lacerations. These strategies include not only the hands-on technique, but also warm compresses, perineal massage, the use of oil or jelly, the Ritgen maneuver and a new perineal protection device. The review by Aasheim reported a decreased risk of third- and fourth-degree lacerations in the perineal massage group (two studies, RR 0.52, 95% CI 0.29 to 0.94).4 This review also showed a similar reduction in third- and fourth-degree lacerations with warm compresses (two studies, RR 0.48, 95% CI 0.28 to 0.84), but no significant changes with use of a Ritgen maneuver. Additional reviews have evaluated delayed versus immediate pushing, with no significant difference in perineal trauma.

Regarding how the interventions may work, initially the hands-on technique was hypothesized to control the velocity of the crowning process and therefore decrease perineal trauma. Given the fact that the hands-on approach has been found to be possibly associated with more perineal lacerations instead of less, some have proposed that the harm may be caused by the hands-on approach's additional pressure resulting in some perineal ischemia. Moreover, using one intervention (e.g. hands-on) may predispose to use other interventions (e.g. episiotomy), which have themselves been proven to increase perineal trauma.

Perhaps a combination of perineal interventions, such as massage or compresses, with a hands-off approach and avoidance of episiotomy, will prove to show improved perineal outcomes. Larger studies, including evaluation specific for nulliparous subjects, are required to make definitive recommendations for management.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestations
* Low risk pregnancies
* 37 to 42 weeks of gestations

Exclusion Criteria:

* Multiple gestations
* Preterm birth

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 70 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Perineal laceration - any degree | at the time of delivery

SECONDARY OUTCOMES:
Incidence of Episiotomy | at the time of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Naples, Italy

IPD SHARING:
Plan to Share IPD: No
none planned

REFERENCES:
- [Derived] Trama U, Bernardi FF, Colacurci D, Saccone G, Guida M. Hands-on vs hands-off technique at the time of delivery and postpartum pelvic floor morbidity: a secondary analysis of a randomized clinical trial. Am J Obstet Gynecol MFM. 2024 Jul;6(7):101383. doi: 10.1016/j.ajogmf.2024.101383. Epub 2024 May 21. No abstract available. PMID 38782091
- [Derived] Califano G, Saccone G, Diana B, Colla Ruvolo C, Ioffredo D, Nappi C, Annella A, Gragnano E, Guida M, Zullo F, Locci M. Hands-on vs hands-off technique for the prevention of perineal injury: a randomized clinical trial. Am J Obstet Gynecol MFM. 2022 Sep;4(5):100675. doi: 10.1016/j.ajogmf.2022.100675. Epub 2022 Jun 10. PMID 35697297